CLINICAL TRIAL: NCT06489938
Title: Effect of Mirror Therapy Combined With Task- vs. Impairment-oriented Rehabilitation Program in Individuals With Stroke
Brief Title: Mirror Therapy Combined With Task- vs. Impairment-oriented Rehabilitation Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I-Shou University (Other)
Responsible Party: Principal Investigator, Yi-chun Li, Neuro-Rehabilitation Research Laboratory (NRRL), I-Shou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISU-OT-Li-01
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Cardiovascular Diseases; Stroke; Cerebrovascular Disorders
Keywords: Rehabilitation; Mirror Therapy
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Cerebrovascular Disorders | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mirror therapy combined with the task-oriented approach (MTT) (Experimental): Each participant will receive the mirror therapy combined with the task-oriented approach 90 minutes daily, three days per week for six weeks.
  Interventions: Behavioral: Mirror therapy; Behavioral: Task-oriented approach
- Mirror therapy combined with the impairment-oriented approach (MTI) (Experimental): Each participant will receive the mirror therapy combined with the impairment-oriented approach 90 minutes daily, three days per week for six weeks.
  Interventions: Behavioral: Mirror therapy; Behavioral: Impairment-oriented approach
- Task-oriented rehabilitation program combined with impairment-oriented rehabilitation program (TI) (Active Comparator): Each participant will receive the task-oriented rehabilitation program combined with the impairment-oriented rehabilitation program 90 minutes daily, three days per week for six weeks.
  Interventions: Behavioral: Task-oriented approach; Behavioral: Impairment-oriented approach

INTERVENTIONS:
Behavioral: Mirror therapy — In mirror therapy, a wooden mirror (41×50×33 cm3) will be positioned in the participant's sagittal midplane, blocking the participant's view of the affected arm performance. We will also provide a foldable bed tray table to ensure that the participants focus on the mirror reflection of the less affected arm. The mirror therapy will consist of movement and functional practices.
  Arms: Mirror therapy combined with the impairment-oriented approach (MTI); Mirror therapy combined with the task-oriented approach (MTT)
Behavioral: Task-oriented approach — The task-oriented approach will provide both bimanual common-goal and dual-goal tasks for the participants.
  Arms: Mirror therapy combined with the task-oriented approach (MTT); Task-oriented rehabilitation program combined with impairment-oriented rehabilitation program (TI)
Behavioral: Impairment-oriented approach — The impairment-oriented approach will focus on the movement components. Arm BASIS or Arm Ability training will be provided based on the severity of the participant's impairment.
  Arms: Mirror therapy combined with the impairment-oriented approach (MTI); Task-oriented rehabilitation program combined with impairment-oriented rehabilitation program (TI)

SUMMARY:
The goal of this clinical trial is to examine the effects of mirror therapy combined with task- vs. Impairment-oriented rehabilitation programs as novel hybrid approaches in individuals with stroke. Participants will receive mirror therapy combined with the task-oriented rehabilitation program (MTT), mirror therapy combined with the impairment-oriented rehabilitation program (MTI), or task-oriented rehabilitation program combined with the impairment-oriented rehabilitation program (TI) 90 minutes per day, three days per week, for six weeks.

ELIGIBILITY:
Inclusion Criteria:

1. A first-ever unilateral stroke ≥3 months
2. Age between 20 and 80 years
3. Baseline Fugl-Meyer Assessment Upper Extremity (FMA-UE) score >10
4. No severe spasticity in any joints of the affected arm
5. Ability to follow the instructions
6. No participation in other studies during the study period
7. Willingness to provide informed written consent.

Exclusion Criteria:

1. Serious medical problems or poor physical conditions that might be detrimental to study participation.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | Baseline, six weeks, and 3 months after completing the intervention
  A standardized tool for evaluating motor impairment for stroke
Revised Nottingham Sensory Assessment | Baseline, six weeks, and 3 months after completing the intervention
  A standardized tool for evaluating sensory impairment for stroke
Chedoke Arm and Hand Activity Inventory | Baseline, six weeks, and 3 months after completing the intervention
  An assessment for bilateral functional abilities
Wolf Motor Function Test | Baseline, six weeks, and 3 months after completing the intervention
  An assessment for both unilateral and bilateral functional abilities

SECONDARY OUTCOMES:
Grip and pinch power | Baseline, six weeks, and 3 months after completing the intervention
  The measurements of the strength of hand movements
Box and block test | Baseline, six weeks, and 3 months after completing the intervention
  A measurement for evaluating functional hand use by measuring the number of blocks moved within a set time
Ten-meter walk test | Baseline, six weeks, and 3 months after completing the intervention
  A test for measuring walking speed and stride length over a fixed distance to assess mobility and functional status
Berg Balance Scale | Baseline, six weeks, and 3 months after completing the intervention
  A measurement for evaluating balance abilities through a series of functional tasks
Motor Activity Log | Baseline, six weeks, and 3 months after completing the intervention
  A self-report tool used to assess the amount and quality of use of an affected limb during daily activities
ABILHAND Questionnaire | Baseline, six weeks, and 3 months after completing the intervention
  A self-reported assessment tool used to measure manual ability by evaluating their perceived difficulty in performing bimanual tasks
Functional independent measure | Baseline, six weeks, and 3 months after completing the intervention
  An assessment tool that evaluates a person's level of disability and functional independence in performing daily activities, covering areas such as self-care, mobility, communication, and social cognition
Nottingham Extended Activities of Daily Living Scale | Baseline, six weeks, and 3 months after completing the intervention
  An assessment tool designed to measure a person's ability to perform daily activities
Stoke Impact Scale | Baseline, six weeks, and 3 months after completing the intervention
  A comprehensive self-reported questionnaire that assesses the impact of a stroke on life
Stroke Self-Efficacy Questionnaire | Baseline, six weeks, and 3 months after completing the intervention
  A tool used to evaluate a stroke survivor's confidence to perform daily activities
Stroke-Specific Measure of Adherence to Home-based Exercises | Six weeks
  A questionnaire designed to assess how consistently stroke participations follow prescribed home programs

CONTACTS AND LOCATIONS:
Overall Officials: Yi-chun Li, Doctor, Principal Investigator — I-Shou University

IPD SHARING:
Plan to Share IPD: No